CLINICAL TRIAL: NCT03877432
Title: Non-invasive Nerve Stimulation for Inhibition of Bladder Incontinence in Spinal Cord Injured Subjects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201605025
Record Dates: First submitted 2019-03-04; First posted 2019-03-15 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dermatome stimulation (Experimental): Check the effect of improving the function of bladder storage and bladder capacity before and after dermatome stimulation.
  Interventions: Device: Dermatome stimulation

INTERVENTIONS:
Device: Dermatome stimulation — Dermatome (S2-S4) stimulation is aimed at improving the function of bladder storage and bladder capacity. A total of 8 serial cystometrograms will be performed: 2 control fills, followed by 4 fills with stimulation, followed by 2 control fills. The minimum (or threshold) stimulation amplitude (T) necessary to elicit the genito-anal reflex was first determined for each subject. Subsequently, each subject received a randomized sequence of cystometric fill trials with and without continuous dermatome stimulation. The dermatome stimulation was randomly stimulated at stimulation amplitudes of 1, 2, 3, and 4 T.

SUMMARY:
Investigators will test S2-S4 dermatome stimulation with spinal cord injury (SCI) individuals using intermittent catheterization to estimate the clinical impact on bladder capacity and continence. For individuals with SCI using intermittent catheterization, investigators hypothesize that dermatome stimulation will decrease bladder spasm frequency and intensity, and reduce bladder incontinence chronically. The goal of this study is to provide objective evidence for the assertion that dermatome stimulation chronically decreases bladder activity and therefore the unwanted side effects of neurogenic bladder. This project will improve the understanding of the neurophysiology of afferent-mediated neural pathways that affect bladder function, and translate recent advances discovered in animal and human studies into clinical research and treatment. The ability to void safely and effectively by electrical stimulation without cutting sacral nerves or the external urethral sphincter would be a major advance. A socially acceptable, predictable and reliable device for reducing incontinence would be widely used and improve quality of life.

DETAILED DESCRIPTION:
Investigators will test S2-S4 dermatome stimulation with SCI individuals using intermittent catheterization to estimate the clinical impact on bladder capacity and continence.

For individuals with SCI using intermittent catheterization, investigators will verify that S2-S4 dermatome stimulation is acutely effective at reducing hyper-reflexive bladder activity during bladder filling. Investigators hypothesize that S2-S4 dermatome stimulation will reduce the number and severity of incontinent episodes, increase bladder capacity, and increase the volume catheterized. By comparing the extended outcomes to the acute laboratory outcomes obtained by ourselves and others, investigators can assess the feasibility of acute urodynamics to identify subjects for implanted devices or future studies.

For individuals with SCI using intermittent catheterization, investigators hypothesize that dermatome stimulation will decrease bladder spasm frequency and intensity, and reduce bladder incontinence chronically. The goal of this study is to provide objective evidence for the assertion that dermatome stimulation decreases bladder activity and therefore the unwanted side effects of neurogenic bladder. These experiments will demonstrate the neurophysiologic response of acute stimulation through urodynamic test, and will also provide increased evidence for future clinical trials through proof of lessened bladder pressures - an important cause of vesico-ureteral reflux and renal injury.

There is a potentially larger population of persons with incomplete SCI than complete SCI who retain sensation in the pelvis who could gain benefit from dermatome stimulation. To examine the outcomes following incomplete SCI (in persons who retain sensation in the pelvis), investigators will test dermatome stimulation to determine the tolerable and effective electrical stimulation parameters in persons that have some degree of preserved motor or sensory function through the lowest sacral spinal cord segments. Investigators will acutely measure the effects of dermatome stimulation on bladder pressure and hyper-reflexic bladder contractions during bladder filling. Investigators hypothesize that dermatome stimulation will increase bladder capacity at stimulus amplitudes that are acutely tolerable to subjects with incomplete SCI. It will determine the feasibility of a non-invasive screening procedure to identify potential candidates for future device implantation, thereby providing a pathway for translation of the technology to implantation.

This project will improve the understanding of the neurophysiology of afferent-mediated neural pathways that affect bladder function, and translate recent advances discovered in animal and human studies into clinical research and treatment. The ability to void safely and effectively by electrical stimulation without cutting sacral nerves or the external urethral sphincter would be a major advance. A socially acceptable, predictable and reliable device for reducing incontinence would be widely used and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Suprasacral SCI
* Neurologically stable
* Skeletally mature, over 18 years of age.
* At least six (6) months post SCI
* Able to understand and comply with study requirements
* Able to understand and give informed consent.

Exclusion Criteria:

* Active sepsis
* Open wound or pressure sores on cutaneous area
* Significant trauma, erosion or stricture of the urethra
* Pregnancy
* Individuals who can not speak.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2021-08-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Wei Peng, Ph.D., Principal Investigator — Professor, School of Biomedical Engineering, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dermatome Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dermatome Stimulation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 10

OUTCOME MEASURES:

1. Primary Outcome: The Changes of Bladder Capacity (mL) by Using Urodynamic Measurement
Description: Investigator will verify that S2-S4 dermatome nerve stimulation is acutely effective at reducing hyper-reflexic bladder activity during bladder filling in urodynamic measurement. All experimental trials will be completed in one day for each subject.
  Serial cystometrograms will be conducted by filling the bladder with saline and recording the volume in the bladder with or without concomitant nerve stimulation.
  A total of 8 serial cystometrograms will be performed: 2 control fills, followed by 4 fills with stimulation, followed by 2 control fills. Stimulation threshold will be randomly given (1-4 folds of stimulation threshold).
  Data from each of 4 stimulation fills per threshold or a total of 4 control fills were averaged. The averaged values are presented per Arm/Group below.
  The interval between every fill is 20-40 min. Investigator will compare the difference of bladder capacity (mL) between giving-control fill and fill with stimulation through statistical analysis.
Time Frame: The outcome measure will be assessed in day 1.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Control: Subjects first received a control fill without genital nerve stimulation (GNS) to determine their bladder capacity (baseline).
- 1T (Threshold): Subjects received 1 fold of stimulation threshold (1T) amplitude while cystometrogram performed.
- 2T (Threshold): Subjects received 2 folds of stimulation threshold (2T) amplitude while cystometrogram performed.
- 3T (Threshold): Subjects received 3 folds of stimulation threshold (3T) amplitude while cystometrogram performed.
- 4T (Threshold): Subjects received 4 folds of stimulation threshold (4T) amplitude while cystometrogram performed.
Arm/Group | Control | 1T (Threshold) | 2T (Threshold) | 3T (Threshold) | 4T (Threshold)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 4
ml | 253 (112) | 346 (116) | 332 (137) | 390 (157) | 401 (134)
Statistical Analysis 1: Comparison: Control vs 1T (Threshold); All data were presented as means ± standard deviations (SDs). Analysis of variance (ANOVA) was used to compare the effects of 1T stimulation amplitude changes on bladder capacity; Test type: Superiority; p = 0.012, ANOVA
Statistical Analysis 2: Comparison: Control vs 2T (Threshold); All data were presented as means ± standard deviations (SDs). Analysis of variance (ANOVA) was used to compare the effects of 2T stimulation amplitude changes on bladder capacity; Test type: Superiority; p = 0.017, ANOVA
Statistical Analysis 3: Comparison: Control vs 3T (Threshold); All data were presented as means ± standard deviations (SDs). Analysis of variance (ANOVA) was used to compare the effects of 3T stimulation amplitude changes on bladder capacity; Test type: Superiority; p = 0.003, ANOVA
Statistical Analysis 4: Comparison: Control vs 4T (Threshold); All data were presented as means ± standard deviations (SDs). Analysis of variance (ANOVA) was used to compare the effects of 4T stimulation amplitude changes on bladder capacity; Test type: Superiority; p = 0.004, ANOVA

2. Secondary Outcome: The Changes of Bladder Pressure (cmH2O) During Urodynamic Measurement
Description: Investigator will verify that S2-S4 dermatome nerve stimulation is acutely effective at reducing hyper-reflexic bladder activity during bladder filling in urodynamic measurement. All experimental trials will be completed in one day for each subject. Serial cystometrograms will be conducted by filling the bladder with saline and recording the pressure in the bladder with or without concomitant nerve stimulation. A total of 8 serial cystometrograms will be performed: 2 control fills, followed by 4 fills with stimulation, followed by 2 control fills. Stimulation threshold will be randomly given (1-4 folds of stimulation threshold). The interval between every fill is 20-40 min. Investigator will compare the difference of bladder capacity (mL) between giving-control fill and fill with stimulation through statistical analysis.
Time Frame: The outcome measure will be assessed in day 1.
Reporting Status: Not Posted, anticipated posting 2021-12

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dermatome Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03877432/Prot_SAP_000.pdf